CLINICAL TRIAL: NCT04556045
Title: Exercise Therapy and Radiation Therapy (EXERT) for Metastatic Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE8821
Record Dates: First submitted 2020-07-28; First posted 2020-09-21 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Malignant Neoplasm of Prostate
Keywords: Exercise; Radiation; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiation Therapy + Exercise Therapy (Experimental): This group will receive exercise intervention in addition to their standard of care radiation treatment. At the baseline visit, they will meet with the certified exercise trainer (CET) and will be provided with a personalized exercise prescription and log to record what they do in between daily radiation treatment visits. The participant will also undergo an in-person exercise session prior to radiation therapy, which will take place either on the same day that the physical function tests are preformed or on a separate day. Participants will exercise between 1 and 7 times/week depending on the patient's tolerance to the exercise prescription. The CET will meet with the participant at every radiation treatment visit for an exercise counseling check-in. After five radiation treatments, the CET will follow-up with the participants via phone call once per week for 4 weeks during the follow-up period.
  Interventions: Behavioral: Exercise therapy
- Radiation Therapy (No Intervention): The observational group will continue with their usual standard of care of radiation therapy. The study team will provide patients with an educational pamphlet at the end of their baseline visit. They will also be provided with a self-directed exercise program framework. Additionally, the participant's medical record will be reviewed for serious adverse events during their time on study. Baseline and final measurements will be obtained.

INTERVENTIONS:
Behavioral: Exercise therapy — The exercise therapy intervention will last 4 weeks. Each participant assigned to this intervention will receive a personalized ET regimen, including in-person, supervised exercise sessions; other activities to be followed at home. Participants will exercise between one and seven times per week depending on their tolerance to the treatment and exercise program.
  Arms: Radiation Therapy + Exercise Therapy

SUMMARY:
This study is being done to determine if patients receiving personalized exercise therapy (versus those who do not receive personalized exercise therapy) have improved quality of life and physical functioning after completing their radiation therapy. Second, the study is being done to find if the quality of life changes during therapy correlate with measurements of inflammation in the blood. Third, the study is being done to see if adding exercise therapy to radiation therapy will improve survival.

DETAILED DESCRIPTION:
In 2018, 30,000 patients were diagnosed metastatic prostate cancer in the US. Short-course radiation therapy (RT) is a mainstay of treatment for symptomatic metastases, and it stimulates an immune response against the tumor. However, RT also decreases systemic interleukin-1 receptor antagonist (IL-1Ra), placing the body in a pro-inflammatory state, and increasing fatigue and reducing quality of life (QOL). Fatigue and QOL are surrogates of the limited 2-20 month survival time. If fatigue and quality of life are improved, then toxicity and survival will follow.

Our long-term goal is to identify the potential for exercise therapy (ET) to improve RT treatment toxicities and outcomes among men diagnosed with metastatic prostate cancer metastatic to distant sites or regional lymph nodes. The mechanistic hypothesis is that adding ET training to RT decreases long-term systemic inflammation, mitigating toxicity thereby widening the therapeutic window.

Objective 1. Quantify the potential of Exercise Therapy (ET) to mitigate Radiation Treatment (RT) toxicities and physical function decline. The hypothesis is that ET mitigates patient-reported quality of life (QOL) and toxicities of RT. Our approach will be to use standardized questionnaires and assessment tools to assess QOL and physical function.

Objective 2. Characterize the immunologic mechanism by which ET mitigates RT toxicity. The hypothesis is that ET mitigates the toxicity of RT (measured in objective 1) by increasing serum interleukin-1Ra (IL-1Ra).

Objective 3. Evaluate the ability of ET to improve survival. Since physical function is a surrogate of survival, the hypothesis is that adding ET to RT will improve overall survival, measured from the date of start of radiotherapy until death.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have lymph node positive or metastatic disease consistent with prostate cancer
* Males ≥18 years of age receiving RT
* Patient receiving 5 fractions or stereotactic body radiation therapy (SBRT)
* Patient may have received prior hormone therapy. Prior or current use of chemotherapy agents is allowed, but not necessary.
* Fluent in written and spoken English
* Must be able to provide and understand informed consent
* Must have an ECOG Performance Status (PS) of ≤ 3
* Primary attending radiation oncologist approval

Exclusion Criteria:

* Performing > 90 minutes/week of exercise therapy prior at time of enrollment
* Evidence in the medical record of an absolute contraindication for exercise
* Cardiac exclusion criteria:
* Class II, III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
* History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty or stenting within the past 6 months prior to the start of radiation therapy
* Uncontrolled arrhythmias; patients with rate-controlled atrial fibrillation for >1 month prior to start of radiation therapy may be eligible
* syncope
* acute myocarditis, pericarditis, or endocarditis
* acute pulmonary embolus or pulmonary infarction
* thrombosis of lower extremities
* suspected dissecting aneurysm
* pulmonary edema
* respiratory failure
* acute non-cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise
* Mental impairment leading to inability to complete study requirements
* In-patient receiving radiation therapy for a radiation emergency (e.g. cord compression, Superior vena cava (SVC) syndrome, brain metastases)
* High risk of fracture or spine instability (Mirels score ≥7, SINS ≥7)
* Children (the protocol will only include men age 18 and older)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life using the Patient-Reported Outcomes Measurement Information System (PROMIS Scale v1.2-Global Health) | At 12 week follow up
  Patient Reported Outcome Measurement Information System (PROMIS) Global Health v1. 2 short form is a 10-item instrument representing multiple domains. Scores are assigned for both Global Physical Health component and Global Mental Health component. The response scores range from 1-5, where 1 = always and 5 = Never. A higher score from responses indicate better health.

SECONDARY OUTCOMES:
Progression free survival | Within 5 years
  The hypothesis is that adding exercise therapy (ET) to radiation therapy (RT) will improve progression free survival, measured using RECIST criteria
Overall survival | Within 5 years
  The hypothesis is that adding exercise therapy (ET) to radiation therapy (RT) will improve overall survival, from the date of start of palliative radiotherapy until death.
Physical Function: Short Physical Performance Battery | At 1 month follow up
  Objectively-measured physical function will be assessed using the Short Physical Performance Battery (SPPB).
  The SPPB is an accumulation of balance tests, 4-meter gait speed, and 5-chair stands. Based on the time needed to complete the chair stands, a score is given. A summation of scores from all tests is taken, ranging from 0 -12. A higher score = Higher physical function.
Aerobic Capacity: Six Minute Walk Test | At 1 month follow up
  Objectively-measured physical function will be assessed using the Six Minute Walk Test (6MWT).
  Distance walked during 6 minutes (measured in meters) is measured. Longer distance = higher aerobic capacity.
Strength: Hand Grip Strength measured by the grip strength dynamometer test | At 1 month follow up
  Reliable and valid evaluation of hand strength can provide an objective index of general upper body strength. Hand grip strength can be quantified by measuring the amount of static force that the hand can squeeze around a dynamometer. The force is measured in kilograms and/or pounds and corresponds.
Health-related Quality of Life: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30, version 3.0) | At 1 month follow up
  QoL will be assessed with the validated 30-item self-assessment questionnaire of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30, version 3.0).
Evaluation of symptomatic toxicity in study participants using the Common Terminology Criteria for Adverse Events- Patient Reported Outcomes (CTCAE-PRO) | At 1 month follow up
  The PRO-CTCAE characterizes the frequency, severity, interference, and presence/absence of symptomatic toxicities that include pain, fatigue, nausea, and cutaneous side effects that can be meaningfully reported from the patient perspective. PRO-CTCAE responses are scored from 0 to 4 (or 0/1 for absent/present) and evaluate the symptom attributes of frequency, severity, interference, amount, presence/absence. Each symptomatic Adverse Event is assessed by 1-3 attributes. Criteria for grading on the CTCAE scale vary by toxicity. Grade 1: asymptomatic or mild symptoms not requiring intervention. Grade 2: moderate symptoms that interfere somewhat with daily function and where some intervention may be indicated. Grade 3: severe symptoms that interfere with daily activities or require more significant intervention. Grade 4: toxicity that is life-threatening, with urgent intervention indicated.
Godin Physical Activity Questionnaire | At 1 month follow up
  Physical activity behavior in the domains of commuting activity, leisure time activities such as cycling, walking, and sports, household and occupational activity will be assessed via a standardized and validated questionnaire, the Godin Physical Activity Questionnaire. Total weekly leisure activity is calculated in arbitrary units by summing the products of the separate components, as shown in the following formula:
  Weekly leisure activity score = (9 × Strenuous) + (5 × Moderate) + (3 × Light) Higher activity score = more active
Fatigue: Fatigue Symptom Inventory | At 1 month follow up
  The Fatigue Symptom Inventory (FSI) assesses the frequency and severity of fatigue as well as its perceived disruptiveness. Frequency is measured as the number of days in the past week (0-7) respondents felt fatigued as well as the percentage of each day on average they felt fatigued (0 = none, 10 = entire day).
Quantification of IL-1Ra in blood | At 1 month follow up
  A 2-4mL blood sample will be collected to determine participants levels of the biomarker IL-1Ra. Samples will be run via ELISA and concentrations will be reported as pg/mL.

OTHER OUTCOMES:
Work Productivity and Activity Impairment Questionnaire | At 1 month follow up
  The Work Productivity and Activity Impairment Questionnaire assesses the effect of patient's health problems on their ability to work and perform regular activities. Subjects self reports as "fill in blank" answers to questions and also as circling a number on a 10 point scale where 0 = Problem had no effect on my work and 10 = Problem completely prevented me from doing my daily activities.
Barriers to Exercise RM 5-FM | At 1 month follow up
  Examines factors that have an impact on the development and implementation of and adherence to a personal physical activity plan. Questions are scored on a range of 0-3 where, Very Unlikely = 0 and Very Likely = 3. Barriers to physical activity fall into one or more of seven categories: lack of time, social influences, lack of energy, lack of willpower, fear of injury, lack of skill, and lack of resources. A score of 5 or above in any category shows that this is an important barrier to overcome.
Exploratory pro-inflammatory (IL-1B, IL-6, TNF-α, IL-8, IL-15, CRP) and anti-inflammatory (IL-10) markers | At 1 month follow up
  A 2-4mL blood sample will be collected to determine participants levels of pro- and anti-inflammatory biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Zaorsky, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share all collected data relevant to results in publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code